CLINICAL TRIAL: NCT03005691
Title: Central Sensitization in Chronic Whiplash Patients: Metabolite Concentrations in the Anterior Cingulate Cortex and Periacueductal Gray Matter
Brief Title: Central Sensitization in Chronic Whiplash Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Other Study IDs: GFSM-HNP
Record Dates: First submitted 2016-12-15; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Pain
Keywords: metabolite; central sensitization; whiplash
MeSH Terms: conditions — Chronic Pain; Whiplash Injuries | interventions — Spectrum Analysis; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Whiplash-Pain: Subjects with chronic whiplash syndrome and pain. The inclusion criteria for pain include the presence of daily pain during the previous 8 weeks. Specifically, pain will be diagnosed based on the pain intensity measured on the 0 to 10 numerical rating scale. The minimum will be 2 points. Subjects will be recruited between the 4 months until 2 years after the whiplash.
  Interventions: Radiation: Spectroscopy; Other: Questionnaires; Procedure: Conditioned Pain Modulation
- Whiplash-no Pain: Subjects with chronic whiplash syndrome and pain. The inclusion criteria for pain include the ausence of daily pain during the previous 8 weeks. Specifically, pain will be diagnosed based on the pain intensity measured on the 0 to 10 numerical rating scale. The maximun will be 2 points. Subjects will be recruited between the 4 months until 2 years after the whiplash.
  Interventions: Radiation: Spectroscopy; Other: Questionnaires; Procedure: Conditioned Pain Modulation
- Non-injured: Subjects without whiplash syndrome. The inclusion criteria are defined as a absence of previous or actual symptoms or signs of neck pain.
  Interventions: Radiation: Spectroscopy; Other: Questionnaires; Procedure: Conditioned Pain Modulation

INTERVENTIONS:
Radiation: Spectroscopy — Spectroscopy is a noninvasive method to assess brain chemistry. The signal of the hydrogen atom attached to a certain molecule or metabolite has a particular frequency associated with a given metabolite. The utility of Spectroscopy is based on the fact thet the nuclei of atoms have magnetic properties that can be used to obtain chemical information regarding both the type of molecule and it is concentration.
  The subjects will be scanned on a 3-T Siemens system and an 12-channel phased-array coil will be used to provide an optimum signal-to-noise ratio for spectroscopy data.
Other: Questionnaires — Questionnaires are important to assess the chronic pain and their impact in the quality of life. For this reason, we will assess the Brief Pain Inventory (BPI), it is used to evaluate the subject's perception of pain severity and its interference. Moreover, we will assess neuropathic pain symptoms with the NPSI to detect paresthesia/dysaesthesia, evoked pain and paroxysmal pain. The catastrophizing score will be measured with the Pain Catastrophizing Helplessness Subscale. Also,we will assess the disability after whiplash using the Neck Disability Index.
Procedure: Conditioned Pain Modulation — Conditioned Pain Modulation over the tenar eminence. The test will be a heat tonic stimulus which evoke a 3-pain intensity. The conditioning stimulus will be a cold water immersion (12ºC)

SUMMARY:
The purpose of this study is to determine whether the metabolite concentrations within the anterior cingulate cortex and periaqueductal gray matter predict the intensity and interference of neuropathic pain after the development of chronic whiplash syndrome.

DETAILED DESCRIPTION:
Persistent chronic pain is a common symptom of whiplash leading to reduced quality of life. Little information is available regarding changes in brain processing areas and change in central sensitization to noxious input during the chronic phase of whiplash. Metabolite concentrations in the anterior cingulate cortex and periaqueductal gray matter may be predictors of neuropathic pain and these changes may explain the development of central sensitization in people with chronic whiplash.

Until now, there is not any study that show this approach.

ELIGIBILITY:
Inclusion Criteria:

* Whiplash syndrome
* Chronic pain
* Age between 18 to 65 years
* 4 months to 2 years after the whiplash syndrome

Exclusion Criteria:

* Neurological disease
* Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered whiplash syndrome. By one hand, patients with chronic pain (minimun 8 weeks) and 2 points or more of pain intensity. By the other hand, patiens without pain (2 points or less of pain intensity).
  By last, subjects without whiplash syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Metabolite concentrations | Baseline at 0 min
  The metabolite concentrations will be measured by magnetic resonance (spectroscopy)
Conditioned Pain Modulation | Baseline at 0 min
  Conditioned Pain Modulation will be measured by a Pathway system (Medoc Ltd)
Brief Pain Inventory | Baseline at 0 min
  Brief Pain Inventory (BPI), it is used to evaluate the subject's perception of pain severity and its interference.
Neurophatic Pain Symptoms Inventory | Baseline at 0 min
  Neurophatic Pain Symptoms Inventory (NPSI), it is used to detect paresthesia/dysaesthesia, evoked pain and paroxysmal pain.
Pain Catastrophizing Helplessness Subscale | Baseline at 0 min
  Pain Catastrophizing Helplessness Subscale it is used to assess the catastrophizing score
Neck Disability Index | Baseline at 0 min
  Neck Disability Index (NDI), it is used to assess the disability after whiplash syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Diego Serrano-Muñoz, MsC, Principal Investigator — Hospital Nacional de Parapléjicos, Toledo

IPD SHARING:
Plan to Share IPD: Yes
To publish in impact journals